CLINICAL TRIAL: NCT06779448
Title: The Effect of Rubber Dam on Objective and Subjective Parameters of Stress During Dental Treatment in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ebru KUCUKYİLMAZ, PROFESSOR, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024/0242
Record Dates: First submitted 2024-12-04; First posted 2025-01-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Dental Anxiety; Dental Fear; Rubberdam; Anesthesia, Dental; Dental Pain
Keywords: dental anxiety; local anesthesia; topical anesthesia; rubber dam; cotton roll; dental stress; stress parameters
MeSH Terms: conditions — Toothache | interventions — Dentists

STUDY DESIGN:
Intervention Model Description: randomized, controlled, single-blinded, split mouth clinical study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- local anesthesia (Active Comparator): local anesthesia application before rubber dam isolation
  Interventions: Other: Evaluation of objective and subjective stress parameters caused by local anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by topical anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by the application of rubber dam during treatments in the patient and dentist; Other: Evaluation of the objective and subjective stress parameters caused by the application of cotton rolls during treatments in the patient and dentist
- topical anesthesia (Active Comparator): topical anesthesia application before rubber dam isolation
  Interventions: Other: Evaluation of objective and subjective stress parameters caused by local anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by topical anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by the application of rubber dam during treatments in the patient and dentist; Other: Evaluation of the objective and subjective stress parameters caused by the application of cotton rolls during treatments in the patient and dentist
- rubber dam (Active Comparator): Rubber dam isolation and evaluation of the associated objective and subjective stress parameters
  Interventions: Other: Evaluation of objective and subjective stress parameters caused by local anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by topical anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by the application of rubber dam during treatments in the patient and dentist; Other: Evaluation of the objective and subjective stress parameters caused by the application of cotton rolls during treatments in the patient and dentist
- cotton roll (Active Comparator): cotton roll insulation and evaluation of the associated objective and subjective stress parameters
  Interventions: Other: Evaluation of objective and subjective stress parameters caused by local anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by topical anesthesia during treatments; Other: Evaluation of objective and subjective stress parameters caused by the application of rubber dam during treatments in the patient and dentist; Other: Evaluation of the objective and subjective stress parameters caused by the application of cotton rolls during treatments in the patient and dentist

INTERVENTIONS:
Other: Evaluation of objective and subjective stress parameters caused by local anesthesia during treatments — Patients were divided according to the randomization procedure. infiltration anesthesia (Maxicaine Forte, Artikain, VEM Drug, Turkey) was performed with a 20-gauge needle. Following the administration of anesthetic, an appropriate size rubber dam and metal clamp was placed i and pit and fissure sealant was applied. The stress parameters of the subjects were recorded at three measurement points. At the conclusion of the treatment, pain perception was evaluated subjectively using the WBFPRS and VAS.
Other: Evaluation of objective and subjective stress parameters caused by topical anesthesia during treatments — Patients were divided i according to the randomization procedure. The topical anesthetic agent (EMLA, AstraZeneca, Cotia, São Paulo, Brazil) was applied using a disposable dental Q-tip for 10-20 seconds. Following the administration of anesthetic, an appropriate size rubber dam and metal clamp was placed i and pit and fissure sealant was applied. The stress parameters of the subjects were recorded at three measurement points. At the conclusion of the treatment, pain perception was evaluated subjectively using the WBFPRS and VAS.
Other: Evaluation of objective and subjective stress parameters caused by the application of rubber dam during treatments in the patient and dentist — Patients were divided into 4 subgroups according to the randomization procedure: topical anesthesia and infiltrative anesthesia before the placement of the clamp and also cotton roll application other side of the arch. The topical anesthetic agent (EMLA, AstraZeneca, Cotia, São Paulo, Brazil) was applied using a disposable dental Q-tip for 10-20 seconds and infiltration anesthesia (Maxicaine Forte, Artikain, VEM Drug, Turkey) was performed with a 20-gauge needle. Following the administration of anesthetics, an appropriate size rubber dam and metal clamp was placed in the mandibular arch, and pit and fissure sealant was applied to the opposite arch. The stress parameters of the subjects and dentist were recorded at three measurement points. At the conclusion of the treatment, pain perception was evaluated subjectively using the WBFPRS and VAS.
Other: Evaluation of the objective and subjective stress parameters caused by the application of cotton rolls during treatments in the patient and dentist — Patients were divided into 4 subgroups according to the randomization procedure: topical anesthesia and infiltrative anesthesia before the placement of the clamp and also cotton roll application other side of the arch. The topical anesthetic agent (EMLA, AstraZeneca, Cotia, São Paulo, Brazil) was applied using a disposable dental Q-tip for 10-20 seconds and infiltration anesthesia (Maxicaine Forte, Artikain, VEM Drug, Turkey) was performed with a 20-gauge needle. Following the administration of anesthetics, an appropriate size rubber dam and metal clamp was placed in the mandibular arch, and pit and fissure sealant was applied to the opposite arch. The stress parameters of the subjects and dentist were recorded at three measurement points. At the conclusion of the treatment, pain perception was evaluated subjectively using the WBFPRS and VAS.

SUMMARY:
Although rubber dam application provides many advantages, several pediatric dentists avoid using it, arguing that it may increase stress for young patients.

The purpose of this clinical study was to evaluate the effect of rubber dam on the subjective and objective stress in children and the effects of preferred anesthesia methods during use of the rubber dam on the same parameters.

A total of 100 children, aged 6-12 years old participated in this study. The selected site of the patients divided cotton roll and rubber dam application group, and the rubber dam group divided also two subgroups as topical and infiltration anesthesia application. Objective parameters of stress of the patients and pulse rate of the operator were measured at three different time points. Pain perception was also evaluated subjectively. The data were statistically analyzed (p<0.05).

DETAILED DESCRIPTION:
This randomized, controlled, single-blinded study included 100 healthy, cooperative children (Frankl Scale, Rating 3-4) aged 6-12 years, classified as ASA I (american assossiation of anesthesiologist), with bilateral fully erupted mandibular first permanent molars requiring pit and fissure sealant procedures. The inclusion criteria were based on the International Caries Detection and Assessment System II, including deep and retentive pits and fissures, no restorations, and no evidence of carious lesions.

The study was planned as split mouth design: For each patient, one tooth was selected for rubber dam isolation, while the corresponding tooth from the opposite quadrant was chosen for cotton roll isolation. The Rubber dam application group divided also into two groups as topical EMLA application, and infiltration anesthesia application. Randomization was performed using manually generated sealed envelopes containing information about which isolation method and anesthesia technique would be used on which side of the jaw (right or left). Random numbers were written on separate papers, folded, and placed in opaque sealed envelopes. Each participant chose an envelope and was assigned the printed participant number. Each number identified the teeth included in the study, the isolation technique specified for each tooth, and the anesthesia method to be used during the rubber dam application. Objective stress parameters (pulse rate, systolic blood pressure and diastolic blood pressure) for the children and the pulse rate of the operator were recorded at three different points: immediately after sitting in the treatment chair and prior to the beginning of the treatment (T1), after light curing of the fissure sealant with cotton roll isolation (T2), and following the completion of treatment and removal of the cotton rolls. Systolic and diastolic blood pressure were measured using an automatic blood pressure monitor (OMRON M2, Omron Healthcare Co., Kyoto, Japan). Pulse rate was evaluated with a fingertip pulse oximeter (LYG88 Pulse Oximeter, China). The operator's pulse rate was also recorded. Pain perception was assessed subjectively post-procedure using the Wong-Baker FACES Pain Rating Scale (WBFPRS) and Visual Analogue Scale (VAS). One week later, the patient was invited to a second appointment for the treatment of the corresponding tooth from the opposite side. At this stage, the teeth were cleaned like in cotton roll group, and the patients were divided into two groups according to the randomization procedure: topical anesthesia and infiltrative anesthesia before the placement of the clamp. The topical anesthetic agent (EMLA, AstraZeneca, Cotia, São Paulo, Brazil) was applied using a disposable dental Q-tip for 10-20 seconds and infiltration anesthesia (Maxicaine Forte, Artikain, VEM Drug, Turkey) was performed with a 20-gauge needle. Following the administration of anesthetics, an appropriate size rubber dam and metal clamp was placed in the mandibular arch, and pit and fissure sealant was applied to the opposite arch. The stress parameters of the subjects were recorded at three measurement points. At the conclusion of the treatment, pain perception was evaluated subjectively using the WBFPRS and VAS.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years child,
* classified as ASA I (american assossiation of anesthesiologist)
* cooperative children
* child with bilateral fully erupted mandibular first permanent molars requiring pit and fissure sealant procedures.

Exclusion Criteria:

* patients/guardians who do not meet the inclusion criteria
* patients/guardians who do not agree to participate in the study.
* child with chronic systemic disease
* non-cooperative children

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
blood pressure | one week intervals about observation/treatment sessions (total time is 2 weeks)
  systolic blood pressure and diastolic blood pressure for the children recorded. Systolic and diastolic blood pressure were measured using an automatic blood pressure monitor (mmHg). (min 20 mmHg- max 320 mmHg) The mean values and standard deviations of these measured values be taken into account.
pulse rate | one week intervals about observation/treatment sessions (total time is 2 weeks)
  pulse rate for the children and the operator recorded. Pulse rate was evaluated with a fingertip pulse oximeter (unit per minute) (min 60- max 160). The mean values and standard deviations of these measured values be taken into account.

SECONDARY OUTCOMES:
pain perception | one week intervals about observation/treatment sessions (total time is 2 weeks)
  Pain perception assessed subjectively post-procedure using the Wong-Baker FACES Pain Rating Scale (WBFPRS). The aforementioned assessments conducted through the assignment of scores. Wong-baker (WBFPRS) is realised as scoring from facial expressions. The lowest score selected from 6 different and graded facial expressions gives the lowest anxiety value (min 0- max 6).
pain perception | one week intervals about observation/treatment sessions (total time is 2 weeks)
  Pain perception is going to assess subjectively post-procedure using the Visual Analogue Scale (VAS). The aforementioned assessments conducted through the assignment of scores. VAS takes values ranging from 0-10 and higher values indicate an increase in patients pain perception. 0 is indicated no pain and 10 is indicated worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA OZDEMIR, RES ASİST, Principal Investigator — İZMİR KATIP CELEBI UNİVERSİTY
Locations (1):
- İzmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
due to concerns about the security of unpublished data

REFERENCES:
- [Background] Ammann P, Kolb A, Lussi A, Seemann R. Influence of rubber dam on objective and subjective parameters of stress during dental treatment of children and adolescents - a randomized controlled clinical pilot study. Int J Paediatr Dent. 2013 Mar;23(2):110-5. doi: 10.1111/j.1365-263X.2012.01232.x. Epub 2012 Mar 8. PMID 22404253
- [Background] Afshari E, Sabbagh S, Khorakian F, Sarraf Shirazi A, Akbarzadeh Baghban A. Reducing pain and discomfort associated with rubber dam clamp placement in children and adolescents: a systematic review and meta-analysis of effectiveness. BMC Oral Health. 2023 Jun 16;23(1):398. doi: 10.1186/s12903-023-03115-7. PMID 37328861
- [Background] Wang Y, Li C, Yuan H, Wong MC, Zou J, Shi Z, Zhou X. Rubber dam isolation for restorative treatment in dental patients. Cochrane Database Syst Rev. 2016 Sep 20;9(9):CD009858. doi: 10.1002/14651858.CD009858.pub2. PMID 27648846
- [Derived] Kucukyilmaz E, Ozdemir T, Savas S. The effect of rubber dam on objective and subjective parameters of stress during dental treatment in children: a randomized clinical trial. BMC Oral Health. 2025 May 30;25(1):855. doi: 10.1186/s12903-025-06250-5. PMID 40448060

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT06779448/Prot_SAP_000.pdf